CLINICAL TRIAL: NCT07321600
Title: The Effects of Resisted Inspiratory Muscle Training Applied in Addition to PSSE-Schroth Exercises on Clinical Outcomes in Individuals With Adolescent Idiopathic Scoliosis.
Brief Title: Resisted Inspiratory Muscle Training Applied in Addition to PSSE-Schroth Exercises
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner KARARTI, Assoc. Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20251223
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Adolescence Idiopathic Scoliosis
Keywords: Schroth; Physiotherapeutic scoliosis-specific exercises; Inspiratory muscle training; Adolescent Idiopathic Scoliosis; 3D motion analysis; plantar pressure; PSSE

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group randomized controlled trial comparing PSSE-Schroth plus resistance inspiratory muscle training versus PSSE-Schroth alone. Interventions will be delivered for 8 weeks, 3 sessions/week (total 24 sessions).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an assessor blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSSE-Schroth + Resistance IMT (Experimental): PSSE-Schroth session will last approximately 45-60 minutes. Exercises will be personalized (by the therapist) according to the individual's curve pattern; emphasis will be placed on the principles of auto-elongation, rotational angular breathing (RAB), derotation, stabilization, and symmetry. Positions will include semi-hanging, prone-on-knees, prone-on-stool, side-lying-on-T-side, side-lying-on-L-side, and supine-tension-with-poles.
  In addition to PSSE-Schroth exercises, resistance IMT will be applied. Training will be conducted using a threshold-loaded IMT device, maintaining Schroth postural alignment. The program will last eight weeks; three days a week, concurrently with PSSE sessions, each session lasting approximately 15-20 minutes.
  Interventions: Other: Physiotherapeutic scoliosis-specific exercises (PSSE-Schroth); Other: PSSE-Schroth + Resistance IMT
- PSSE-Schroth (Active Comparator): Participants will receive PSSE-Schroth exercises alone for 8 weeks, 3 sessions/week (24 sessions). PSSE-Schroth session will last approximately 45-60 minutes. Exercises will be personalized (by the therapist) according to the individual's curve pattern; emphasis will be placed on the principles of auto-elongation, rotational angular breathing (RAB), derotation, stabilization, and symmetry. Positions will include semi-hanging, prone-on-knees, prone-on-stool, side-lying-on-T-side, side-lying-on-L-side, and supine-tension-with-poles.
  Interventions: Other: Physiotherapeutic scoliosis-specific exercises (PSSE-Schroth)

INTERVENTIONS:
Other: Physiotherapeutic scoliosis-specific exercises (PSSE-Schroth) — Participants will perform a standardized PSSE-Schroth exercise program under supervision. Sessions will be delivered three times per week for 8 weeks (total 24 sessions). Exercises will be individualized according to scoliosis pattern and clinical assessment
  Other Names: Schroth exercises; PSSE
Other: PSSE-Schroth + Resistance IMT — Participants will receive threshold-loaded inspiratory muscle training in addition to PSSE-Schroth. IMT will be supervised and performed three times per week for 8 weeks, aligned with the exercise sessions. Training will be progressed according to individual tolerance and protocol targets
  Other Names: Resistance IMT
  Arms: PSSE-Schroth + Resistance IMT

SUMMARY:
This prospective randomized controlled trial will evaluate whether adding resisted inspiratory muscle training (IMT) to Physiotherapeutic Scoliosis-Specific Exercises (PSSE)-Schroth exercises provides additional benefits on clinical outcomes in individuals with adolescent idiopathic scoliosis. Participants will be randomly assigned to either PSSE-Schroth plus IMT or PSSE-Schroth alone. Both groups will receive supervised exercise sessions three times per week for 8 weeks (24 sessions). Outcomes will be assessed before and after the intervention and will include clinical measures (e.g., Cobb angle, angle of trunk rotation, Posterior Trunk Symmetry Index, The Walter Reed Visual Assessment Scale), respiratory muscle performance (maximal inspiratory pressure/maximal expiratory pressure, six-minute walk test) and related physiological parameters, functional performance (balance, 3D kinematics, plantar pressure analysis, isokinetic strength), sleep quality, and health-related quality of life (Scoliosis Research Society- 22, Italian Spine Youth Quality of Life). The study is expected to enroll approximately 45 participants.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity that may adversely affect thoracic volume, respiratory mechanics, postural symmetry, balance, functional capacity, and health-related quality of life. While physiotherapeutic scoliosis-specific exercises (PSSE), including the Schroth method, have demonstrated clinical benefit, the evidence regarding the added value of integrating structured inspiratory muscle training (IMT) with PSSE remains limited, particularly in studies using comprehensive physiological and biomechanical outcome sets.

This prospective, randomized controlled trial will investigate whether adding resisted IMT to a standardized PSSE-Schroth program provides additional improvements in clinical outcomes in adolescents with AIS.

Eligible participants will be females aged 10-18 years diagnosed with AIS, with Cobb angle between 10° and 45°, angle trunk rotation (ATR) ≥5°, and skeletal immaturity criteria consistent with Risser ≤3 and Sanders ≤4. Participants with non-idiopathic scoliosis, recent spine surgery/major trauma, contraindications to exercise, relevant systemic/neurological conditions, or recent participation in PSSE/IMT programs will be excluded.

Participants will be randomly allocated to one of two groups: (1) PSSE-Schroth plus resistance IMT or (2) PSSE-Schroth alone. Both groups will receive supervised sessions for 8 weeks, three times per week (total 24 sessions). The independent variable is the exercise protocol, and dependent variables include clinical measures.

The trial aims to provide a multidimensional evaluation of the potential additive effects of IMT when integrated with PSSE-Schroth, offering clinically relevant evidence to refine conservative rehabilitation strategies for AIS.

ELIGIBILITY:
Inclusion Criteria:

Female adolescents aged 10-18 years.

Diagnosis of adolescent idiopathic scoliosis (AIS).

Cobb angle between 10° and 45°.

Angle trunk rotation (ATR) ≥ 5°.

Risser ≤ 3 and Sanders ≤ 4.

No scoliosis-related procedure within the last 6 months.

No contraindication to exercise.

Exclusion Criteria:

Non-idiopathic scoliosis (neuromuscular, congenital, syndromic).

Inability to achieve ≥80% adherence/compliance.

History of spinal surgery or major trauma.

Cardiopulmonary diseases contraindicating exercise.

Neurological, rheumatological, vestibular, or systemic diseases.

Acute musculoskeletal injury or impaired skin integrity.

Participation in a regular PSSE-Schroth or IMT program within the last 3 months.

Intellectual disability or communication difficulties preventing protocol adherence.

Newly initiated brace treatment or high risk of non-compliance with brace management.

Lack of informed consent.

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-12-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test | Baseline and after 8 weeks (24 supervised sessions).
  The Six-Minute Walk Test (6MWT) is a tool designed to assess functional exercise capacity, with a particular focus on individuals suffering from cardiopulmonary conditions. The distance walked in six minutes on a flat, straight course, typically 30 metres long, is recorded. The distance measured reflects submaximal exercise capacity. The 6MWT is a valuable tool in the assessment of disease progression, the evaluation of rehabilitation outcomes, and the determination of treatment response.
Change in Cobb Angle | Baseline and after 8 weeks (24 supervised sessions).
  Cobb angle will be measured on standard standing posteroanterior radiographs. The primary outcome is the change in Cobb angle from baseline to post-intervention.
Respiratory muscle strength - maximal inspiratory pressure (MIP) | Baseline and Week 8 (end of 24 supervised sessions).
  Maximal inspiratory pressure (cmH₂O) will be measured using a digital manometer. The primary outcome is the change in MIP from baseline to after the 8-week intervention, and the between-group difference in this change (PSSE-Schroth + resistance IMT vs PSSE-Schroth alone).

SECONDARY OUTCOMES:
Angle of Trunk Rotation (ATR) | Baseline and immediately after the 8-week intervention (24 sessions)
  Angle of trunk rotation will be measured using a Bunnell scoliometer during the forward bend test. The outcome will be reported as change from baseline to post-intervention and compared between groups.
Posterior Trunk Symmetry Index (POTSI) | Baseline and immediately after the 8-week intervention.
  Posterior trunk symmetry will be evaluated using the Posterior Trunk Symmetry Index (POTSI). Change from baseline to post-intervention will be analyzed to assess the effect of adding inspiratory muscle training to PSSE-Schroth.
Walter Reed Visual Assessment Scale - Turkish version (WRVAS-TR) | Baseline and Week 8
  Perceived trunk deformity will be assessed with the Turkish version of the Walter Reed Visual Assessment Scale (WRVAS-TR). The outcome will be the change in total score from baseline to after the intervention.
Health-related Quality of Life - SRS-22 | Baseline and Week 8
  Health-related quality of life will be assessed using the Scoliosis Research Society-22 questionnaire. The outcome will be the change in total and domain scores from baseline to after the intervention.
Health-related Quality of Life - ISYQOL | Baseline and Week 8
  Health-related quality of life will be assessed using the Italian Spine Youth Quality of Life (ISYQOL) questionnaire. Change in total score from baseline to after the 8-week intervention will be analyzed.
Sleep quality (Pittsburgh Sleep Quality Index) | Baseline and Week 8
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The outcome will be the change in PSQI global score from baseline to after the intervention.
Daytime sleepiness (Epworth Sleepiness Scale) | Baseline and Week 8
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (adult or child/adolescent version, as appropriate). The outcome will be the change in total score from baseline to after the 8-week intervention and comparison between groups.
Trunk muscle activation (surface EMG) | Baseline and Week 8
  Trunk muscle activation patterns will be evaluated using surface electromyography (sEMG) from selected trunk muscles during standardized postural or functional tasks. The outcome will be the change in normalized EMG activity from baseline to after the 8-week intervention
Spinal and pelvic kinematics (3D motion analysis) | Baseline and Week 8
  Three-dimensional motion analysis will be used to quantify spinal and pelvic kinematics during standardized tasks. The outcome will be the change in relevant kinematic parameters from baseline to after the 8-week intervention.
Plantar pressure distribution (baropodometric analysis) | Baseline and Week 8
  Plantar pressure distribution and load symmetry will be assessed using a baropodometric platform. The outcome will be the change in plantar pressure variables (e.g., forefoot-rearfoot loading and left-right symmetry) from baseline to after the 8-week intervention.
Knee muscle strength (isokinetic quadriceps and hamstrings) | Baseline and Week 8
  Knee extensor (quadriceps) and flexor (hamstring) muscle strength will be measured using an isokinetic dynamometer during concentric knee flexion and extension. The outcome will be the change in peak torque (normalized to body mass) from baseline to after the 8-week intervention.
Postural Control Assessment | Baseline and after 8 weeks (24 supervised sessions).
  Individuals' postural control in static-eyes open, static-eyes closed, and dynamic positions will be measured using the Korebalance® System. The Korebalance® System is a computerised platform that combines balance assessment with exercise, providing a technologically advanced solution for balance-related concerns.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to participant privacy considerations and the inclusion of minors.